CLINICAL TRIAL: NCT07188623
Title: VR-Enhanced BA for Older Adults With Major Depressive Disorder
Brief Title: Virtual Reality-Enhanced Behavioral Activation for Older Adults With Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Margot Paul, PsyD, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-80275
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Depression - Major Depressive Disorder; Older Adults (65 Years and Older); Behavioral Activation Treatment; Virtual Reality Therapy
Keywords: Depression; Older adult; major depressive disorder; MDD; behavioral activation; VR; virtual reality; older adults
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-Enhanced BA (Experimental): Participants will perform all of their behavioral activation in virtual reality (VR). Participants will meet with the clinician once a week for four weeks (5 sessions). In between weekly therapy sessions, participants will be asked to pick at least one pleasurable activity to enjoy in VR per day. Participants will complete their post-VR surveys and add and schedule activities on separate worksheets.
  Interventions: Behavioral: VR-Enhanced BA

INTERVENTIONS:
Behavioral: VR-Enhanced BA — Participants will choose at least one "activity" per day to complete in the loaned HTC VIVE Flow Immersive Glasses extended reality over the course of the week. These activities are chosen from the headset and include video 360.

SUMMARY:
The primary aims of this study are to assess the feasibility, acceptability, and tolerability of using an immersive virtual reality (VR) headset to engage in behavioral activation (BA) for older adults diagnosed with major depressive disorder (MDD). The secondary aim of this study is to explore the efficacy of using VR to enhance BA therapy in a clinical MDD older adult population.

DETAILED DESCRIPTION:
This research study is looking for older adults with depression to participate in a research study on the use of virtual reality (VR)-enhanced behavioral activation therapy for depression. The purpose of the study is to learn more about using VR to enhance behavioral activation as a treatment for MDD.

Behavioral activation is defined as identifying pleasant and/or mastery activities, scheduling them into your calendar, and completing the identified activities during the week. The identification of pleasant and mastery activities will begin in session with a therapist and will include tracking the participant's hourly activities with the activity/ mood monitoring form and identifying how much pleasure and/or mastery the participant may feel when completing these activities. The following session, the participant and therapist will be able to identify patterns and discuss how to decrease unhelpful behaviors and explore the participant's interests and values to increase positive behaviors. The clinician will explain how to use the loaned VR headset, which looks similar to glasses. The participant will be asked to choose VR activities of interest to complete in between sessions and schedule them into their activity scheduling sheet. They will be asked to rate their mood before and after engaging with the VR headset. A discussion of barriers to completion and problem-solving will also be discussed in session. Once per week, the participant will also be asked to complete a post-VR questionnaire which will ask questions about presence felt in the headset, any physical discomfort while in the headset, and their feelings about the headset. During the last session, treatment and skills will be reviewed and the participant will be asked to provide verbal feedback.

ELIGIBILITY:
Inclusion Criteria:

* Patient must meet DSM V criteria for MDD
* Patient must be at least 65 years of age
* Patient must be English speaking
* Without cognitive impairment

Exclusion Criteria:

* Substance Use Disorders in past year
* Any psychosis or bipolar I disorder
* Any seizure in the last 6 months or untreated epilepsy
* Current nonsuicidal self-injury or parasuicidal behavior
* Current suicidal urges and intent
* Changing psychotherapy treatment within three months of study entry
* Changing psychotropic medication(s) within two months of study entry

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Depression Scores on the GDS-15 From Baseline to Session 5 | Assessed at the beginning of sessions 1, 2, 3, 4, and 5 (days 1, 8, 15, 22, and 29)
  How participants' depression scores on the Geriatric Depression Scale (GDS-15) change over time using VR-enhanced BA. The GDS-15 is a 15-question screener with a score range of 0-15, with 15 indicating the most severe depression and 0 indicating a lack of depression symptoms. The greater the change over time, the greater the symptom reduction.

SECONDARY OUTCOMES:
Participant's Desire to Continue Using Virtual Reality (VR) After the Study Ends | Assessed after session 5, at the end of week 4.
  This outcome was measured using the "Intention to use Technology " questions of the Technology Acceptance Model questionnaire. These are questions 11, 12, and 13 and allow participants the option of circling Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), or Strongly Agree (4). With 3 questions, the total range was 0-12 (higher scores indicate greater acceptance).
Participant's Satisfaction With the VR-Enhanced BA Treatment | Assessed after session 5, at the end of week 4
  This outcome was measured using the "Attitudes Toward Use " questions of the Technology Acceptance Model questionnaire. These are questions 7, 8, 9, and 10 and allow participants the option of circling Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), or Strongly Agree (4). With 4 questions, the total range was 0-16 (higher scores indicate greater acceptance).
Participant's Use of the VR Headset | Assessed after session 5, at the end of week 4.
  This was measured by noting the amount of times the XR headset is used during the 4-week study period.
Participant's Acceptance of VR-Enhanced BA Treatment | Assessed after session 5, at the end of week 4.
  This was measured using the overall Technology Acceptance Model questionnaire, which encompasses 13 questions and allows participants the option of circling Strongly Disagree (0), Disagree (1), Neutral (2), Agree (3), or Strongly Agree (4), yielding a range of 0-52 (higher scores indicate greater acceptance).
How Well Can Participants Tolerate the VR-Enhanced BA Treatment? | Assessed after session 5, at the end of week 4.
  This was determined by the Simulator Sickness Questionnaire, which names 16 adverse symptoms and asks participants to circle as compared to baseline: No more than usual (0), Slightly more than usual (1), Moderately more than usual (2), or Severely more than usual (3), yielding a range of 0-48 (lower scores indicate greater tolerability).
How Present Did Individuals in the VR-Enhanced BA Treatment Feel in the Headset? | Assessed after session 5, at the end of week 4.
  This was measured using the Presence Questionnaire, which asks three questions and asks the participants to circle either Not at all (0), Slightly (1), Moderately (2), Strongly (3), or Very Strongly (4), yielding a range of 0-12 (higher scores indicate greater presence).

CONTACTS AND LOCATIONS:
Overall Officials: Margot Paul, PsyD, Principal Investigator — Stanford University; Kim Bullock, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No